CLINICAL TRIAL: NCT03515213
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of Fenofibrate as a Treatment for Huntington's Disease
Brief Title: Safety and Efficacy of Fenofibrate as a Treatment for Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Leslie Thompson, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20163022
Record Dates: First submitted 2017-08-02; First posted 2018-05-03 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Drug: Fenofibrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenofibrate — 145mg of fenofibrate
  Arms: Active
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to study the safety and efficacy of fenofibrate, an FDA-approved drug for high cholesterol and/or elevated triglycerides (fats), as a treatment for Huntington's disease (HD). Subjects who meet the entry criteria will be randomized (3:1) to either 145mg of fenofibrate or placebo.

ELIGIBILITY:
Inclusion Criteria:

* An adult of either sex, ages 25-85 inclusive,
* Have proficiency with written and spoken English and corrected vision or hearing to complete the cognitive testing,
* Are able to give informed consent,
* Have good overall health status with no known problems anticipated over the course of the trial,
* Have a diagnosis of HD supported by positive gene test within the past 6 months.

Exclusion Criteria:

* Other major neurological disease [e.g., multiple sclerosis, parkinson's disease, cortical stroke, etc]
* Clinically significant hepatic or renal disease,
* Current or recent (< 1 month) use of dopamine blocking agents such as tetrabenazine, anticonvulsants, neuroleptics, HAART, antiemetics, and antipsychotics for any reason,
* Current use of Warfarin (Coumadin). Enrollment in another investigational drug study within the prior three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Hermanowicz, MD, Principal Investigator — University of California, Irvine; Leslie Thompson, PhD, Study Director — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Placebo
Started | 9 | 1
Completed | 9 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Ten participants baseline assessments analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 9 | 1 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 1 | 9
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (9.9) | 49.9 | 54.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 1 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 1 | 10
UHDRS TFC [Mean (Standard Deviation); unit: units on a scale] — United Huntington Disease Rating Scale, Total Functional Capacity, greater than or equal to 7 was the inclusion criteria and is a scale representing functional capacity. A higher score represents worsening and lower score represents better functional capacity.
  units on a scale | 9.78 (2.44) | 8 (0) | 9.6 (2.37)

OUTCOME MEASURES:

1. Primary Outcome: Change in PGC-1alpha RNA Expression
Description: Change in PGC-1alpha RNA expression from Baseline, Month 3 and Month 6
Time Frame: Baseline compared to 3 and 6 months.
Population: Fenofibrate vs placebo
Measure: Mean (Standard Deviation); unit: Log 2 fold change
Arm/Group | Active | Placebo
Number analyzed (Participants) | 9 | 1
Log 2 fold change
  Month 3 | -0.02190716 (0.9017336) | 0.3160562
  Month 6 | 0.07414876 (0.4723322) | 0.4800263

2. Primary Outcome: Change in PGC-1alpha Protein Abundance.
Description: Mean change in PGC-1alpha protein abundance.
Time Frame: Baseline compared to 3 and 6 months.
Measure: Mean (Standard Deviation); unit: Log 2 fold change
Arm/Group | Active | Placebo
Number analyzed (Participants) | 9 | 1
Log 2 fold change
  Month 3 | 0.2609123 (1.031904) | -0.02029792
  Month 6 | 0.02375246 (0.9096516) | 0.3185422

3. Secondary Outcome: Change in Fenofibric Acid Level.
Description: Change in Fenofibric acid abundance from Baseline to 3 and 6 months.
Time Frame: Baseline to 3 and 6 months.
Population: Fenofibrate vs placebo
Measure: Mean (Standard Deviation); unit: Ng/ml
Arm/Group | Active | Placebo
Number analyzed (Participants) | 4 | 1
Ng/ml
  Baseline | 64 (117.48) | 5 (0)
  Month 3 | 9037 (7114.1) | 10 (0)
  Month 6 | 10905 (5900.77) | 19 (0)

4. Secondary Outcome: Change in Unified Huntington Disease Rating Scale Motor Score.
Description: Unified Huntington Disease Rating Scale (UHDRS) Motor (total score range 0-124 where higher score = greater impairment)
Time Frame: Baseline and 6 months
Population: Fenofibrate vs placebo. Change in motor scores from baseline to month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 9 | 1
score on a scale
  Baseline | 19.56 (11.87) | 34 (0)
  Month 6 | 21.22 (17.22) | 27 (0)

5. Secondary Outcome: Change in Montreal Cognitive Assesment Score.
Description: Montreal Cognitive Assessment (total score range 0-30, higher score = less impairment)
Time Frame: Baseline compared to 3 and 6 months.
Population: Changes in cognition scores from baseline to month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 9 | 1
score on a scale
  Baseline | 24.222 (3.701) | 18
  Month 3 | 25.778 (3.866) | 16
  Month 6 | 25.667 (4.093) | 22

6. Secondary Outcome: Changes in Unified Huntington Disease Rating Scale - Behavioral
Description: Unified Huntington Disease Rating Scale (UHDRS) Behavioral Scale (total score range 0-100 where 100 = 100% independent)
Time Frame: Baseline, Month 3 and 6 months
Population: Changes in independence assessment scores from baseline, month 3 to month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 9 | 1
score on a scale
  Baseline | 9.778 (2.438) | 8
  Month 3 | 8.333 (3.674) | 9
  Month 6 | 8.444 (3.575) | 8

7. Secondary Outcome: Change in Functional Assessment Scores
Description: Clinical Global Impression (CGI-I); (total score range 1-7 where higher score = greater impairment), and Unified Huntington Disease Rating Scale (UHDRS) Total Functional Capacity Assessment ( total score range 0-13, higher score = less impairment)
Time Frame: Baseline compared to 3 and 6 months.
Population: Change in functional assessment scores from baseline, month 3 to month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 9 | 1
score on a scale
  Baseline | 3.222 (1.09) | 3
  Month 3 | 3.571 (0.787) | 3
  Month 6 | 3.571 (0.787) | 3

ADVERSE EVENTS:
Time Frame: Adverse events data were collected over 6 months.
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed, but no adverse events were observed over 6 months.
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/1
Other Adverse Events (participants affected / at risk) | 0/9 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03515213/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03515213/ICF_001.pdf